CLINICAL TRIAL: NCT00748644
Title: MAINtenance of Remission Using RITuximab in Systemic ANCA-associated Vasculitis
Brief Title: Efficacy Study of Two Treatments in the Remission of Vasculitis
Acronym: MAINRITSAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 070703
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Wegener Granulomatosis; Microscopic Polyangiitis
Keywords: Wegener's granulomatosis,; microscopic polyangiitis,; ANCA-associated vasculitis,; rituximab,; azathioprine
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Rituximab; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Experimental drug = rituximab for maintenance
  Interventions: Drug: Rituximab
- 2 (Active Comparator): Comparator drug = azathioprine for maintenance
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: Rituximab — rituximab infusion will be performed at J1, J15, M6, M12 and M18(i.e. a total of 5 infusions), at the dose of 500 mg at a fixed dosage.
  All patients received corticosteroids, starting from induction with prednisone (or equivalent) at a dose of 1 mg/kg/day with gradual tapering according to a regimen adjusted to body weight over a mean of 18 months since diagnosis.
  Arms: 1
Drug: Azathioprine — azathioprine (2 mg/kg/d) for 12 months, then progressively tapered until its discontinuation at month 22.
  All patients received corticosteroids, starting from induction with prednisone (or equivalent) at a dose of 1 mg/kg/day with gradual tapering according to a regimen adjusted to body weight over a mean of 18 months since diagnosis.
  Arms: 2

SUMMARY:
Study of the efficacy of rituximab for maintenance treatment in systemic ANCA-associated vasculitis: prospective, multicenter, controlled, randomized comparative study of rituximab versus azathioprine

DETAILED DESCRIPTION:
Randomized, controlled, national, multicenter, prospective study to compare between azathioprine (conventional therapy) and rituximab in patients with systemic ANCA-associated vasculitis, in remission (achieved with an induction treatment combining corticosteroids and an immunosuppressant, mainly intravenous pulses of cyclophosphamide, and plasma exchanges and/or polyvalent immunoglobulins when indicated) after the first flare of the disease (new diagnosis) or after a relapse. It is planned to stratify patients by first flare (66% of the patients) or relapse (33% of the patients). Patients complying with the inclusion criteria may be included when they are in remission from their vasculitis. Patients who have already received biologics (antiCD20, antiTNFα) will not be included. Patients will be included at the time of remission and then randomized. They will receive maintenance treatment by azathioprine for 18 months or a rituximab infusion every 6 months until month 18 (i.e. a total of 4 infusions), at the dose of 375 mg/m2 (maximum dosage, 500 mg). ANCA status and CD19+ lymphocyte count will be monitored but will not be used to adjust therapy. After the 18 month length of maintenance phase, i.e. after stopping immunosuppressive maintenance therapy, patients will be followed for an additional 10 month period. Patients with Wegener's granulomatosis will be prescribed cotrimoxazole 160/800 tid (for 2 additional years).

ELIGIBILITY:
Inclusion Criteria:

* Wegener's granulomatosis Or microscopic polyangiitis complying Or kidney-limited disease With or without detectable ANCA (anti-neutrophil cytoplasmic antibodies) at the time of diagnosis or relapse, and at remission.
* Who have achieved remission using a treatment combining corticosteroids and an immunosuppressive agent according to current French guideline, including corticosteroids, cyclophosphamide IV or oral (the use of another immunosuppressant is allowed, according to the current French guidelines, as well as plasma exchanges and/or IV immunoglobulins).
* Interval of 1 month between the end of the immunosuppressant treatment and the randomization time
* Age > 18 years and < 75 years when the diagnosis is confirmed.
* Informed and having signed the consent form to take part in the study.

Exclusion Criteria:

* Other systemic vasculitis
* Secondary vasculitis (following neoplastic disease or an infection in particular)·
* Induction treatment with a regimen not corresponding to that recommended in France.
* Patient who has not achieved remission.·
* Patient who has already received a treatment by biological agents (monoclonal antibody - antiCD20 or antiTNFα).
* Incapacity or refusal to understand or sign the informed consent form.
* Incapacity or refusal to adhere to treatment or perform the follow-up examinations required by the study. Non-compliance·
* Allergy, documented hypersensitivity or contraindication to the study medication (cyclophosphamide, corticosteroids, azathioprine, rituximab),
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
* Patients receiving allopurinol cannot be included if the allopurinol must absolutely be maintained.
* Pregnancy, breastfeeding. Women of childbearing age must use a reliable method of contraception throughout the duration of immunosuppressive treatment up to 1 year after the last infusion of rituximab
* Infection by HIV, HCV or HBV
* Progressive, uncontrolled infection requiring a prolonged treatment (tuberculosis, HIV infection, etc.).
* Severe infection declared during the 3 months before randomization (CMV, HBV, HHV8, HCV, HIV, tuberculosis).
* Progressive cancer or malignant blood disease diagnosed during the 5 years before the diagnosis of vasculitis. Patients suffering from non-metastatic prostate cancer or those cured of a cancer or a malignant blood disorder for more than 5 years and not taking any antineoplastic agents for more than 5 years may be included.
* patients presenting a systemic disease receiving protocolized treatments (azathioprine, rituximab) which could have unexpected and inappropriate side effects.
* Participation in another clinical research protocol during the 4 weeks before inclusion.
* Any medical or psychiatric disorder which, in the investigator's opinion, may prevent the administration of treatment and patient follow-up according to the protocol, and/or which may expose the patient to a too greater risk of an adverse effect.
* No social security
* Churg and Strauss syndrome
* viral, bacterial or fungic or mycobacterial infection uncontrolled in the 4 weeks before the inclusion
* history of deep tissue infection (fasciitis, osteomyelitis, septic arthritis)in the first year before the inclusion
* History of chronic and severe or recurrent infection or history of preexisting disease predisposing to severe infection
* Severe immunodepression
* Administration of live vaccine in the four weeks before inclusion
* severe chronic obstructive pulmonary diseases (VEMS < 50 % or dyspnea grade III)
* chronic heart failure stade III and IV (NYHA)
* History of recent acute coronary syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2008-10; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of major relapse (BVAS>10) in each group at the end of the maintenance treatment (18 months treatment + 10 months follow-up) | 28 months

SECONDARY OUTCOMES:
To assess the number of adverse events and their severity in each group | 28 months
Number of patients with ANCA in each group | 28 months
mortality rate in each group | 28 months
number of minor relapse in each group | 28 months
Cumulated dose and the length of corticosteroid treatment in each group at 28 months | 28 months
same criteria with an analysis at 6 months after the end of maintenance treatment | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Loic Guillevin, MD, PhD, Study Director — French Vasculitis Study Group
Locations (1):
- Hopital Cochin, Paris, France

REFERENCES:
- [Result] Pugnet G, Pagnoux C, Terrier B, Perrodeau E, Puechal X, Karras A, Khouatra C, Aumaitre O, Cohen P, Maurier F, Decaux O, Ninet J, Gobert P, Quemeneur T, Blanchard-Delaunay C, Godmer P, Carron PL, Hatron PY, Limal N, Hamidou M, Ducret M, Daugas E, Papo T, Bonnotte B, Mahr A, Ravaud P, Mouthon L, Guillevin L; French Vasculitis Study Group. Rituximab versus azathioprine for ANCA-associated vasculitis maintenance therapy: impact on global disability and health-related quality of life. Clin Exp Rheumatol. 2016 May-Jun;34(3 Suppl 97):S54-9. Epub 2016 Mar 25. PMID 27049404
- [Result] Guillevin L, Pagnoux C, Karras A, Khouatra C, Aumaitre O, Cohen P, Maurier F, Decaux O, Ninet J, Gobert P, Quemeneur T, Blanchard-Delaunay C, Godmer P, Puechal X, Carron PL, Hatron PY, Limal N, Hamidou M, Ducret M, Daugas E, Papo T, Bonnotte B, Mahr A, Ravaud P, Mouthon L; French Vasculitis Study Group. Rituximab versus azathioprine for maintenance in ANCA-associated vasculitis. N Engl J Med. 2014 Nov 6;371(19):1771-80. doi: 10.1056/NEJMoa1404231. PMID 25372085
- [Derived] Romand X, Paclet MH, Chuong MV, Gaudin P, Pagnoux C, Guillevin L, Terrier B, Baillet A. Serum calprotectin and renal function decline in ANCA-associated vasculitides: a post hoc analysis of MAINRITSAN trial. RMD Open. 2023 Oct;9(4):e003477. doi: 10.1136/rmdopen-2023-003477. PMID 37903568
- [Derived] Terrier B, Pagnoux C, Perrodeau E, Karras A, Khouatra C, Aumaitre O, Cohen P, Decaux O, Desmurs-Clavel H, Maurier F, Gobert P, Quemeneur T, Blanchard-Delaunay C, Bonnotte B, Carron PL, Daugas E, Ducret M, Godmer P, Hamidou M, Lidove O, Limal N, Puechal X, Mouthon L, Ravaud P, Guillevin L; French Vasculitis Study Group. Long-term efficacy of remission-maintenance regimens for ANCA-associated vasculitides. Ann Rheum Dis. 2018 Aug;77(8):1150-1156. doi: 10.1136/annrheumdis-2017-212768. Epub 2018 May 3. PMID 29724729
- See also: Website of the French Vasculitis Study Group — http://www.vascularites.org